CLINICAL TRIAL: NCT04419480
Title: Hemodynamic Monitoring to Prevent Adverse Events foLlowing cardiOgenic Shock Trial
Acronym: HALO-Shock
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U19-05-3608
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Cardiogenic Shock; Heart Failure; Ambulatory Hemodynamic Monitoring
MeSH Terms: conditions — Shock, Cardiogenic; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CardioMEMS Implant Group (Experimental): Following enrollment, patients randomized 1:1 to post-discharge implantation of the CardioMEMS device will receive that device ≤14 days following discharge from the index hospitalization for Cardiogenic Shock, in addition to local standard of care medical therapy.
  Interventions: Device: CardioMEMS implantation with routine ambulatory pulmonary artery pressure monitoring and medication optimization
- Non-CardioMEMS Implant Group (No Intervention): Following enrollment, patients randomized 1:1 to post-discharge standard of care will be treated according to local standard of care medical therapy following their index hospitalization for Cardiogenic Shock.

INTERVENTIONS:
Device: CardioMEMS implantation with routine ambulatory pulmonary artery pressure monitoring and medication optimization — Implantation of CardioMEMS Device in patients following admission for Cardiogenic shock, with regular ambulatory pulmonary artery pressure monitoring and medication optimization for the treatment of heart failure.
  Arms: CardioMEMS Implant Group

SUMMARY:
Pilot Prospective Randomized Unblinded Pragmatic Trial of Pulmonary Artery Hemodynamic Monitoring Following Hospitalization for Cardiogenic Shock

ELIGIBILITY:
Inclusion Criteria:

1. Subject or legal representative has signed Informed Consent Form (ICF) and the patient has the capacity to participate in the study and complete the study questionnaires, in the estimation of the study investigator.
2. Age ≥ 18 years
3. NYHA Class III with dyspnea upon mild physical activity, regardless of left ventricular ejection fraction (LVEF).
4. Survive to discharge during a current hospital admission with cardiogenic shock (CS) as defined by clinical criteria previously used in cardiogenic shock trials: systolic blood pressure < 90 mmHg for > 30 minutes or requiring infusion of catecholamines to maintain the systolic blood pressure above 90 mmHg, with evidence of end-organ dysfunction such as pulmonary edema or impaired end-organ perfusion including altered mentation, oliguria with urine output < 30 mL/h, or serum lactate > 2 mmol/L (5). Hemodynamic criteria include cardiac index ≤ 1.8 L/min/m2 without vasoactive pharmacologic agents, or cardiac index ≤ 2.2 L/min/m2 and pulmonary artery occlusion pressure ≥ 15 mmHg with vasoactive agents.
5. Patients must have internet and phone access (to allow communication of the implanted device with the researchers).

Exclusion Criteria:

1. Technical obstacles which pose an inordinately high procedural risk, in the judgment of the investigator.
2. Treatment with ongoing mechanical circulatory support (MCS) such as a durable left ventricular assist device (LVAD) or recipient of a heart transplantation for the treatment of cardiogenic shock during the index hospitalization for CS.
3. If of childbearing potential with a positive pregnancy test.
4. Transition to hospice care.
5. Intolerance to or inability to adhere to antiplatelet therapy for 1 year after device implantation.
6. Presence of an active, uncontrolled infection.
7. Any condition other than heart failure that could limit survival to less than 6 months
8. Discharge to facility other than acute rehabilitation or to the ambulatory setting.
9. No access to internet or phone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hierarchical primary endpoint | 6 months
  Hierarchical endpoint at 6-months, including death (or mortality-equivalent including left ventricular assist device implantation or heart transplantation), recurrent cardiovascular hospitalization, health related quality of life change from baseline, measured by the Minnesota Living with Heart Failure Questionnaire (MLHFQ) as a continuous score, and change in log-transformed NT-proBNP level from enrollment to 6 months, evaluated by the win ratio according to the Finkelstein-Schoenfeld method

SECONDARY OUTCOMES:
Health related quality of life change from baseline | 2 months and 6 months
  Health related quality of life change from baseline, measured by the Minnesota Living with Heart Failure Questionnaire (MLHFQ) as a continuous score at 2 months and 6 months following admission for CS.hemodynamic monitor is safe in the high-risk CS population.
All-cause mortality | 6 months
  All-cause mortality from enrollment.
All-cause mortality or cardiovascular hospitalization | 6 months
  Time to first all-cause mortality or cardiovascular hospitalization.
All-Cause Hospitalization | 6 months
  Time to all-cause hospitalization.
Unscheduled hospital visits (including Emergency Department and Outpatient Diuretic Infusion Clinic) | 6 months
  Time to all unscheduled hospital visits (including Emergency Department and Outpatient Diuretic Infusion Clinic)
Change in NT-pro-B-type natriuretic peptide (NT-pro-BNP) | 6 months
  Change in NT-pro-B-type natriuretic peptide (NT-pro-BNP) from enrollment to 6 months follow up.
Achieved guideline directed medical therapy for heart failure | 6 months
  Achieved guideline directed medical therapy for heart failure with reduced ejection fraction at 6 months, measured by achievement of >50% of the guideline targeted optimal dosing of angiotensin receptor blocker or angiotensin converting enzyme inhibitor or angiotensin receptor neprilysin inhibitor, beta-blocker, and mineralocorticoid receptor antagonist.
Safety of early post-discharge implantation of a pulmonary artery hemodynamic monitoring. | 6 months
  Safety of early post-discharge implantation of a pulmonary artery hemodynamic monitor in the high-risk CS population, including device-related or system-related complications or pressure-sensor failures.

CONTACTS AND LOCATIONS:
Overall Officials: Shashank Sinha, MD MSc, Principal Investigator — Inova Fairfax Medical Campus
Locations (1):
- Inova Fairfax Medical Campus, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No